CLINICAL TRIAL: NCT04449081
Title: Knowledge, Attitude and Practice About COVID-19 and Awareness of Infection Control to Prevent COVID-19 Transmission in Clinics and Perception About Online Learning During Lock Down Period: A Cross-sectional Study
Brief Title: Knowledge, Attitude and Practice of Dental Students About COVID-19
Status: Completed | Type: Observational
Sponsor: Melaka Manipal Medical College (Other)
Responsible Party: Principal Investigator, Rajesh Hosadurga, Professor, Melaka Manipal Medical College
Other Study IDs: MelakaMMC
Record Dates: First submitted 2020-06-25; First posted 2020-06-26 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Acute Respiratory Distress Syndrome; Corona Virus Infection; Acute Lung Injury; Fever; Myalgia; Cough; Dyspnea; Septic Shock; Bleeding
Keywords: Humans; COVID-19; Online learning; Perception
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections; Acute Lung Injury; Fever; Myalgia; Cough; Dyspnea; Shock, Septic; Hemorrhage; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Knowledge, Attitude, Practice, Awareness, Preference — KAP, Awareness level and Preference were assessed using questionnaires

SUMMARY:
Coronavirus disease 2019 (abbreviated "COVID- 19") is a pandemic respiratory disease that is caused by a novel coronavirus and was first detected in December 2019 in Wuhan, China. The disease is highly infectious, and its main clinical symptoms include fever, dry cough, fatigue, myalgia, and dyspnoea.1 In China, 18.5% of the patients with COVID-19 developed to the severe stage, which is characterized by acute respiratory distress syndrome, septic shock, difficult-to-tackle metabolic acidosis, and bleeding and coagulation dysfunction.

After China, COVID-19 spread across the world and many governments implemented unprecedented measures like suspension of public transportation, the closing of public spaces, close management of communities, and isolation and care for infected people and suspected cases. The Malaysian government had enforced Movement Control Order (MCO) from 18th March to 4th May 2020 and henceforth Conditional Movement Control Order (CMCO) until 9th June 2020. The battle against COVID-19 is still continuing in Malaysia and all over the world.

Due to the CMO and CMCO in the country, public and private universities have activated the e-learning mode for classes and as the government ordered, universities are closed and no face-to-face activities allowed. This has forced students of all disciplines including dentistry to stay at home which are wide-spread across Malaysia and shift to e- learning mode. To guarantee the final success for fight against COVID-19, regardless of their education status, students' adherence to these control measures are essential, which is largely affected by their knowledge, attitudes, and practices (KAP) towards COVID-19 in accordance with KAP theory. Once the restrictions are eased students have to come back and resume their clinical work in the campus.

Hence, in this study we assessed the Knowledge, Attitude, and Practice (KAP) towards COVID-19 and the students preference for online learning.

DETAILED DESCRIPTION:
Due to the CMO and CMCO in the country, public and private universities have activated the e-learning mode for classes and as the government ordered, universities are closed and no face-to-face activities allowed. This has forced students of all disciplines including dentistry to stay at home which is wide-spread across Malaysia and shift to e-learning mode. To guarantee the final success for the fight against COVID-19, regardless of their education status, students' adherence to these control measures is essential, which is largely affected by their knowledge, attitudes, and practices (KAP) towards COVID-19 in accordance with KAP theory.

Background:

In the KAP study conducted among residents in China, it was noticed that KAP scores were associated with a lower likelihood of negative attitudes and preventive practices towards COVID-2019. Most Chinese residents of a relatively high socioeconomic status, in particular women, are knowledgeable about COVID-19, hold optimistic attitudes, and have appropriate practices towards COVID-19. Health education programs aimed at improving COVID-19 knowledge are helpful for Chinese residents to hold optimistic attitudes and maintain appropriate practices. In a cross-sectional study among pregestational and pregnant women was conducted in Shaanxi, China, women at the periconceptional period in Shaanxi lacked the total KAP level of periconceptional healthcare, especially those who live in rural areas and have less education. The authors concluded that government agencies should reinforce more effective primary preventive measures and policies for the prevention of adverse pregnancy outcomes.

In a study aimed to assess the level of awareness, perception, and attitude regarding COVID-19 and infection control among Jordanian dentists, the authors concluded that Jordanian dentists were aware of COVID-19 symptoms, mode of transmission, and infection controls and measures in dental clinics. But dentists had limited comprehension of the extra precautionary measures that protect the dental staff and other patients from COVID-19. They also recommended that it would be best practice to send National and international guidelines established by the regional and national dental associations to all registered dentists during a crisis, including the COVID-19 pandemic, to ensure that dentists are well informed and aware of best practices and recommended disease management approaches.

The outbreak of COVID-19 was unprecedented and forced many universities to launch online courses to ensure the continuity of teaching-learning activities, with students staying at homes or dorms. It is a massive, challenging shift to move all the existing courses online in a matter of days. In general, a complete online course requires an elaborate lesson plan design, teaching materials such as audio and video contents, as well as technology support teams.

Many academic institutions in Malaysia commit themselves to eLearning because they believe in its effectiveness as an alternative approach to the traditional classroom method of disseminating information. A study conducted on e-learning shows that higher education institutions in Malaysia offer more than 50% of their courses online. The data also shows that 13.8% of lecturers provide more than 80% online learning materials and that 44.6% of students prefer to read materials uploaded by their lecturers. The findings also show that students' preference for online courses is very encouraging. In fact, lecturers also agree that the integration of e-learning into their courses has benefited students. In general, it clearly shows that the application of e-learning is accepted by lecturers and students of HEIs as an effective means of communication.

A national study was conducted to evaluate the self-perceived preparedness of final-year dental undergraduate students in dental public universities in Malaysia. The authors concluded that confidence and experience in some clinical skills, cognitive and behavioral attributes could be improved to facilitate their transition into independent dental practice after graduation. This is best possible in face-to-face teaching. So given this unprecedented situation, it will be best to assess the perception of dental students towards online teaching.

ELIGIBILITY:
Inclusion Criteria:

* All consenting participants of year 3, 4 and undergraduate dental students studying at Faculty of Dentistry, Melaka-Manipal Medical College, Melaka
* Age - 18-30 years
* All gender

Exclusion Criteria:

* Incomplete questionnaires

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All consenting participants of year 3, 4 and undergraduate dental students studying at Faculty of Dentistry, Melaka-Manipal Medical College, Melaka, were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Knowledge, Attitude, Practice of dental students towards COVID-19 | 4 months
  KAP towards COVID-19 was assessed using validated questionnnaire

SECONDARY OUTCOMES:
Awareness level about Infection control to prevent COVID-19 transmission in clinics | 4 months
  Awareness level about Infection control to prevent COVID-19 transmission in clinics was assesed using a standardized questionnaire
Preference towards online learning. | 4 months
  Preference towards online learning. was assessed using a standard questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Hosadurga, Ph.D, Principal Investigator — Melaka-Manipal Medical College, Melaka, Malaysia
Locations (1):
- Faculty of Dentistry, Melaka-Manipal Medical College, Melaka Tengah, Melaka, Malaysia

IPD SHARING:
Plan to Share IPD: No
No personal details of the participant will be shared.

REFERENCES:
- [Background] Zhong BL, Luo W, Li HM, Zhang QQ, Liu XG, Li WT, Li Y. Knowledge, attitudes, and practices towards COVID-19 among Chinese residents during the rapid rise period of the COVID-19 outbreak: a quick online cross-sectional survey. Int J Biol Sci. 2020 Mar 15;16(10):1745-1752. doi: 10.7150/ijbs.45221. eCollection 2020. PMID 32226294
- [Background] Khader Y, Al Nsour M, Al-Batayneh OB, Saadeh R, Bashier H, Alfaqih M, Al-Azzam S, AlShurman BA. Dentists' Awareness, Perception, and Attitude Regarding COVID-19 and Infection Control: Cross-Sectional Study Among Jordanian Dentists. JMIR Public Health Surveill. 2020 Apr 9;6(2):e18798. doi: 10.2196/18798. PMID 32250959
- [Background] Asiry MA. Dental students' perceptions of an online learning. Saudi Dent J. 2017 Oct;29(4):167-170. doi: 10.1016/j.sdentj.2017.03.005. Epub 2017 Aug 2. PMID 29033527